CLINICAL TRIAL: NCT05491447
Title: A Phase 2 Clinical Trial to Evaluate the Safety, Clinical Effects, and Systemic Exposure of a Topical Application of BMX-010 Ointment in Adult Subjects With Atopic Dermatitis
Brief Title: A Clinical Trial of BMX-010 in Adult Subjects With Atopic Dermatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding constraints
Sponsor: BioMimetix JV, LLC (Industry)
Collaborators: Innovaderm Research Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: BMX-DERM-02
Record Dates: First submitted 2022-08-03; First posted 2022-08-08 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Atopic Dermatitis
Keywords: AD
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: Group 1, Group 2
Who Masked: Participant, Outcomes Assessor
Masking Description: Group 1 participation is open-label. For Group 1, subjects who consent to participate in the PK portion of the study will not be randomized and will receive BMX-010.
  Group 2 is partially blinded. The identification of investigational product is done by lot numbers. The subject will be blinded to the treatment arm and efforts will also be made to maintain a blinded clinical center assessor in this clinical trial. This will be done by ensuring the assessor does not handle the investigational product. Additional efforts may be made to protect the study blinding to ensure at minimum the subject and assessor are blinded, and other staff as appropriate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Study Drug Treated, BMX-010 0.5% (Active Comparator): n=72
  Interventions: Drug: BMX-010
- Study Drug Treated, BMX-010 0.1% (Active Comparator): n=72
  Interventions: Drug: BMX-010
- Placebo Treated (Placebo Comparator): n=72
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMX-010 — Ointment
  Arms: Study Drug Treated, BMX-010 0.1%; Study Drug Treated, BMX-010 0.5%
Drug: Placebo — Ointment
  Arms: Placebo Treated

SUMMARY:
Phase 2 clinical trial conducted in 2 parts: Part 1 - Pharmacokinetics and Part 2 - Randomized and Placebo Controlled (subject and clinical assessors will be blinded). Study Product will be applied to AD BID days 1-28. There will be weekly visits from Baseline (day 1) through Day 29. There is a final follow up visit 2 weeks after.

DETAILED DESCRIPTION:
Group 1 is an open-label safety cohort to determine the PK profile of the active study drug, BMX-010 ointment. At least 3 and up to 12 subjects will be enrolled to analyze the safety and pharmacokinetics of BMX-010 ointment. If a subject cannot complete the required PK blood draws, another subject will be enrolled to ensure at least 3 subjects complete the PK blood draws. Subjects will not be randomized and all subjects in this group will be dispensed BMX-010. Dispensing information will be provided by IWRS. Study drug will be administered in clinic on Day 1 and also Day 8 (the first study drug application of the day) in order to obtain pre-dose PK blood draws. Once a minimum of 3 subjects complete all of the PK blood draws (through Day 8) and the data is analyzed, the Clinical Safety Committee (CSC) will review and determine if enrollment to Group 2 can begin.

Enrollment of subjects into Group 2 will not begin until the PK and safety data from a minimum of three subjects enrolled in Group 1 is obtained and analyzed, and proceeding with Group 2 has been approved by the sponsor.

Once enrollment in Group 2 begins, the subjects will be randomized into Arm A, B, or C.

Group 2 is a randomized, partially blinded (where neither the subjects nor the appropriate clinical center staff are told which treatment or intervention participants are receiving), placebo-controlled cohort designed to further test the safety and efficacy of BMX-010 ointment vs. placebo. Up to approximately 216 adult subjects with AD will be enrolled. At the baseline visit, subjects will be randomized to receive BMX-010 (0.5% or 0.1%) or placebo in a 1:1:1 ratio, by a permuted block randomization schema.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age at the time of consent;
* Diagnosis of AD, as defined by the criteria of Hanifin and Rajka, stable in the last 4 weeks, with onset at least 6 months prior to screening (information obtained from medical chart or subject's physician, or directly from the subject).
* Group 1 only: Subjects should have AD covering approximately 2-5% of the BSA at screening and Day 1 (excluding scalp, face, palms, soles, genitals, and folds). Subjects will treat approximately 5% of their BSA (excluding scalp, face palms, soles, genitals, and folds).
* Group 2 only: 4. Group 2 only: Subject has active AD lesions covering 2-25% of the BSA at screening and Day 1 (excluding scalp, face, palms, soles, genitals, and folds from BSA calculation).
* EASI score >/= 5 (greater than or equal to 5) at screening and Day 1.
* vIGA-AD score ≥ 2 (greater than or equal to 2) at screening and Day 1.
* Candidate for topical treatment of AD;
* Subjects must be willing to apply an emollient of their choice during study.
* Females of child-bearing potential must have a negative urine pregnancy test at screening and on the day of the first drug administration;
* Females of child-bearing potential must be willing to use 2 methods of contraception deemed adequate through the trial and for 1 month thereafter to be eligible for, and continue participation in, the study.
* Ability to complete the study in compliance with the protocol, including agreement in writing to apply IP only to the assigned areas.
* Ability to understand and provide written informed consent.

Exclusion Criteria:

* Subjects with AD only located on the hands and feet.
* Subjects with clinically infected AD.
* Subjects for which systemic pharmacotherapy or phototherapy for the treatment of AD is indicated or required.
* Treatment with systemic retinoids, corticosteroids, immunomodulators or immunosuppressive agents (e.g., methotrexate, cyclosporine), cytotoxic agents, interferon, upadacitinib, abrocitinib, or baricitinib within 4 weeks of the Baseline visit or anticipated need for any of these therapies during the study period.
* Treatment with topical corticosteroids, crisaborole, ruxolitinib, Vitamin D analogs, keratolytics, coal tar, calcineurin inhibitors, antihistamines or any other therapeutic agents besides bland emollients within 2 weeks of the Baseline visit or anticipated need for any of these.
* Treatment with a biological agent (such as a monoclonal antibody) within a period of time of 12 weeks or 5 half-lives (whichever is longer) prior to Day 1.
* Subject has used systemic antibiotics within 2 weeks or topical antibiotics within 1 week prior to Day 1. Of note, subjects with herpes labialis or genitalis and use of antivirals for these diseases are allowed.
* Subject has used dupilumab within 26 weeks prior to Day 1.
* Subject has used doxepin within 1 week prior to Day 1.
* Subject has used hydroxyzine or diphenhydramine within 1 week prior to Day 1.
* Subject has used topical products containing urea within 1 week prior to Day 1.
* Subject has used medical devices, and bleach baths within 2 weeks prior to Day 1.
* Subject has had excessive sun exposure, is planning a trip to a sunny climate, or has used tanning booths within 4 weeks prior to Day 1 or is not willing to minimize natural and artificial sunlight exposure during the study. Use of sunscreen products (except on treated lesions) and protective apparel are recommended when sun exposure cannot be avoided.
* Subject has received an intravenous immunoglobulin (IVIg) therapy within 12 weeks prior to Day 1.
* AD triggered by an unavoidable environmental allergen or irritant.
* Contact dermatitis or drug-induced skin reactions.
* Concomitant skin disease that could confound clinical evaluations or increase risk to the subject.
* Systemic or skin infection requiring antimicrobial therapy within 14 days prior to Baseline.
* Systemic chemotherapy or radiotherapy within 4 weeks of the Baseline Visit.
* Immunocompromise of any cause, known human immunodeficiency virus infection, or acquired immunodeficiency syndrome, including patients receiving immune therapy.
* Pregnancy, planned pregnancy, lactation, or inadequate contraception as judged by the investigator.
* Active drug or alcohol dependence.
* Significant acute or chronic medical, neurological, or psychiatric illness that, in the judgment of the investigator, could compromise subject safety, limit the subject's ability to complete the study, and/or compromise the objectives of the study; clinically significant renal or hepatic insufficiency.
* History of malignancy, unless clinically cured for more than 5 years prior to Baseline. This exclusion does not apply to basal and squamous cell carcinomas of skin and carcinoma in situ of the cervix if they have been adequately treated and are clinically judged to be cured.
* Subject had a major surgery within 8 weeks prior to Day 1 or has a major surgery planned during the study.
* Participation in another investigational drug or vaccine trial concurrently or within 4 weeks for nonbiological investigational products or devices or 12 weeks (or 5 half-lives) for biological investigational products prior to Screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2023-01-08 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Eczema Area and Severity Index at Week 4 | 28 days
  Evaluate the change in Eczema Area and Severity Index score in subjects with active AD treating with BMX-010 0.5% and 0.1% ointment compared with vehicle from baseline to week 4.
Incidence of treatment emergent adverse events and changes from baseline in vital signs and clinical laboratory parameters | 28 days
  Compare treatment emergent adverse events, as well as changes from baseline in vital signs and clinical laboratory parameters in subjects with active AD receiving BMX-010 0.5% and 0.1% ointment compared with vehicle.

SECONDARY OUTCOMES:
Change from baseline in Eczema Area and Severity Index at weeks 1, 2, and 3. | 21 days
  Evaluate the change in Eczema Area and Severity Index score subjects with active AD treating with BMX-010 0.5% and 0.1% ointment compared with vehicle at weeks 1, 2, and 3.
Proportion of subjects who achieve Eczema Area and Severity Index-50 and Eczema Area and Severity Index -75 at Weeks 1, 2, 3 and 4. | 28 days
  Eczema Area and Severity Index-50 and Eczema Area and Severity Index-75 measures indicate the proportion of subjects with active AD with improvement over 50% and 75% based on the Eczema Area and Severity Index at weeks 1, 2, 3, and 4 in subjects treating with BMX-010 0.5% and BMX-010 0.1% compared to vehicle .
Change from baseline in Body Surface Area x validated Investigator Global Assessment of Atopic Dermatitis scoreat Weeks 1, 2, 3, and 4 | 28 days
  Evaluate the change in Body Surface Area x validated Investigator Global Assessment of Atopic Dermatitis scores in subjects with active AD treating with BMX-010 0.5% and 0.1% ointment compared with vehicle at weeks 1, 2, 3 and 4.
Change from baseline in body surface area at Weeks 1, 2, 3, and 4. | 28 days
  Evaluate the change in Body Surface Area in subjects with active AD treating with BMX-010 0.5% and 0.1% ointment compared with vehicle at weeks 1, 2, 3 and 4.
Change from baseline in validated Investigator Global Assessment of Atopic Dermatitis at Weeks 1, 2, 3, and 4. | 28 days
  Evaluate the change in validated Investigator Global Assessment of Atopic Dermatitis score in subjects with active AD treating with BMX-010 0.5% and 0.1% ointment compared with vehicle at weeks 1, 2, 3 and 4.
Proportion of subjects who achieve a validated Investigator Global Assessment of Atopic Dermatitis score of Almost clear (1) and/or Clear (0) with a 2-point reduction at Weeks 1, 2, 3, and 4. | 28 days
  Evaluate the proportion of subjects who achieve a validated Investigator Global Assessment of Atopic Dermatitis score of Almost clear (1) and/or Clear (0) with a 2-point reduction at Weeks 1, 2, 3, and 4 in subjects with active AD treating with BMX-010 0.5% and 0.1% ointment compared with vehicle at weeks 1, 2, 3 and 4.
Change from baseline in the Pruritus Numerical Rating Scale (NRS) at Weeks 1, 2, 3, and 4. | 28 days
  Evaluate the change in the Pruritus Numerical Rating Scale score from baseline to weeks 1, 2, 3, and 4 in subjects with active AD treating with BMX-010 0.5% and 0.1% ointment compared with vehicle.
Change from baseline in Modified Pruritus Numerical Rating Scale (Current Itch Intensity; 30 minutes and 4 hours post-dose) on Day 1. | 1 day
  Evaluate the change in Modified Pruritus Numerical Rating Scale (Current Itch Intensity; 30 minutes and 4 hours post-dose) compared to the pre-dose value on Day 1 in subjects with active AD treating with BMX-010 0.5% and 0.1% ointment compared with vehicle.
Measurement of plasma concentrations of BMX-010 in participants receiving active treatment | 8 days
  Pharmacokinetic plasma samples will be collected on Day 1 and Day 8 at pre-dose and 1 and 3 hours post dose to evaluate the systemic exposure profile and pharmacokinetic (PK) behavior of BMX-010 under the conditions of this trial.

OTHER OUTCOMES:
Change and percent change from baseline of subject-reported Patient-Oriented Eczema Measure (POEM) scores to Week 4. | 28 days
  Evaluate the change and percent change in scores of the subject-reported Patient-Oriented Eczema Measure (POEM) scores from baseline to week 4 in subjects with active AD treating with BMX-010 0.5% and 0.1% ointment compared with vehicle.
Change from baseline in answers on the subject reported PRO questions regarding itching at Weeks 1, 2, 3 and 4 | 28 days
  Evaluate the change of subject report Quality of Life questions regarding itching at weeks 1, 2, 3, and 4 in subjects with active AD treating with BMX-010 0.5% and 0.1% ointment compared with vehicle.

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Cahaba Dermatology & Skin Health Center, Birmingham, Alabama
  - Dermatology Trial Associates, Bryant, Arkansas
  - Johnson Dermatology, Fort Smith, Arkansas
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Axon Clinical Research, Inglewood, California
  - Colorado Skin Care, Englewood, Colorado
  - Skin Care Research, Boca Raton, Florida
  - Driven Research LLC, Coral Gables, Florida
  - RM Medical Research, Miami Lakes, Florida
  - Lenus Research, Sweetwater, Florida
  - Physicians Research Group, West Lafayette, Indiana
  - Skin Sciences, Pllc, Louisville, Kentucky
  - Clinical Trials Management, LLC, Mandeville, Louisiana
  - Revival Research Institute, LLC, Troy, Michigan
  - National Allergy and Asthma Research, LLC., North Charleston, South Carolina
  - J&S Studies, Inc., College Station, Texas
  - Austin Institute for Clinical Research, Pflugerville, Texas
  - Jordan Valley Dermatology Center, South Jordan, Utah
  - Dermatology Specialists of Spokane (Dermatology Specialists of Spokane, PLLC), Spokane, Washington

IPD SHARING:
Plan to Share IPD: Undecided